CLINICAL TRIAL: NCT00786682
Title: A Phase II Study of Docetaxel and Modulation of Autophagy With Hydroxychloroquine for Metastatic Hormone Refractory Prostate Cancer
Brief Title: Docetaxel and Hydroxychloroquine in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of improved efficacy compared to historical controls, competing studies
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000617998; P30CA072720 (NIH); CINJ-080805 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel and Hydroxychloroquine (Experimental): Drug: Docetaxel 75 mg/m2 intravenously every 21 days on Day 1 of the treatment cycle
  Drug: hydroxychloroquine 200 mg twice daily
  A cycle is defined as an interval of 21 days.
  Interventions: Drug: docetaxel; Drug: hydroxychloroquine

INTERVENTIONS:
Drug: docetaxel
Drug: hydroxychloroquine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hydroxychloroquine may help docetaxel work better and kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with hydroxychloroquine works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the antitumor activity, in terms of tumor response rate, of docetaxel in combination with hydroxychloroquine in patients with metastatic, hormone-refractory, chemotherapy-naive prostate cancer.

Secondary

* To measure time to disease progression and overall survival.
* To determine the feasibility and safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral hydroxychloroquine twice daily on days 1-21 and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days (up to 6 courses with docetaxel) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Metastatic disease, as demonstrated by bone scan and/or CT scan of the abdomen/pelvis
  * Must demonstrate disease progression after initial hormone therapy (including bicalutamide and flutamide)
  * No prior chemotherapy allowed
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* ANC > 1,500/μL
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm^3
* Serum creatinine < 2.0 mg/dL or creatinine clearance > 50 mL/min
* Total bilirubin normal
* SGOT and/or SGPT < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No second primary malignancy except for most in situ carcinomas (e.g., adequately treated nonmelanoma carcinoma of the skin) or other malignancy treated ≥ 5 years ago with no evidence of recurrence
* No history or symptoms of cardiovascular disease, including any of the following:

  * NYHA class II-IV cardiovacular disease within the past 6 months
  * Coronary artery disease
  * Arrhythmias
  * Conduction defects with risk of cardiovascular instability
  * Uncontrolled hypertension
  * Clinically significant pericardial effusion
  * Congestive heart failure
* No uncontrolled intercurrent illness including ongoing active infection that would limit compliance with study requirements
* No rheumatoid arthritis or systemic lupus erythematosus requiring treatment
* No psoriasis or porphyria
* No known HIV infection
* No hypersensitivity to 4-aminoquinoline compounds, including hydroxychloroquine sulfate, chloroquine phosphate, and amodiaquine
* No retinal or vision changes from prior 4-aminoquinoline compound use
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No known G-6PDH deficiency
* Neurotoxicity ≤ grade 1

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No prior taxane
* At least 4 weeks since prior therapy (including surgery and radiotherapy)
* At least 1 week since prior herbal supplements
* At least 6 weeks since prior bicalutamide
* At least 4 weeks since prior flutamide
* No current hydroxychloroquine for treatment or prophylaxis

  * Prior hydroxychloroquine allowed
* No other concurrent investigational or commercial agents or therapies, including chemotherapy, immunotherapy, hormonal cancer therapy, radiotherapy, surgery for cancer, or experimental therapy
* Concurrent luteinizing-hormone releasing-hormone agonists allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (7):
- United States (7):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Peters University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) and a community hospital in New Jersey, part of the CINJ Oncology Group, from February 2009 through August 2010.
Period: Overall Study
Arm/Group | Docetaxel and Hydroxychloroquine
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Hydroxychloroquine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate - Primary Endpoint is a 50% Decline in PSA or Normalization of PSA.
Description: We will use a two-stage optimal Simon's design with a 5% significance level and 80% power to detect an increase in response rate from 50% to 70%. The first stage will enroll 15 patients. If there are 8 or fewer responses among these 15 patients, we will consider the combination therapy to not be worthy of further study, and stop the trial. If we find 9 or more responses, we will proceed to the second stage, and accrual continues for a total of 43 patients. If we see 26 or fewer responses out of 43, then no further investigation of the drug is warranted. If we see 27 or more responses out of 43, then further investigation of the drug will be considered. The "expected" sample size of the trial is 23.5 with the null response rate of 50%.
Time Frame: 4 years
Population: Upon reviewing response data for the first 8 patients, we noted that there were no responses thus far. As per the two-stage optimal Simon's design, we would need 8 responses in 15 patients to proceed to stage 2 but we would not have crossed that threshold. The study was stopped due to lack of improved efficacy compared to historical controls.
Arm/Group | Docetaxel and Hydroxychloroquine
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Disease Progression
Time Frame: 10 years
Population: Study was terminated prematurely and insufficient data was collected to assess this outcome measure.
Arm/Group | Docetaxel and Hydroxychloroquine
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Time Frame: 10 years
Population: Study was terminated prematurely and insufficient data was collected to assess this outcome measure.
Arm/Group | Docetaxel and Hydroxychloroquine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Docetaxel and Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Hydroxychloroquine (N=11)
Hemorrhage, GU - Bladder (Blood and lymphatic system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Hydroxychloroquine (N=11)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (6)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Pain - Back (General disorders) | 2 (3)
Pain - Joint (General disorders) | 2 (2)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Chest wall (General disorders) | 1 (1)
Pain - Chest/thorax NOS (General disorders) | 1 (1)
Pain - Dental/teeth/peridontal (General disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Pain - Neck (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (7)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1)
Cardiac General (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (3)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1 (1)
Hemorrhage, GU - Urinary NOS (Blood and lymphatic system disorders) | 1 (1)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory ) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes